CLINICAL TRIAL: NCT04739007
Title: Pulmonary Physiologic Assessment of Patients on Veno-arterial Extracorporeal Membrane Oxygenation (VA ECMO)
Status: Withdrawn | Type: Observational
Why Stopped: Not enough personnel to follow the trial- study was withdrawn
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lorenzo Berra, MD, Reginald Jenney Associate Professor of Anaesthesia, Massachusetts General Hospital
Other Study IDs: 2020P003054
Record Dates: First submitted 2021-01-28; First posted 2021-02-04 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Cardiac Arrest; Pulmonary Injury
MeSH Terms: conditions — Heart Arrest; Lung Injury | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Veno-arterial extracorporeal membrane oxygenation (VA-ECMO) — VA-ECMO used for resuscitation after cardiac arrest
Device: Electrical Impedance Tomography (EIT) — EIT used to demonstrate ventilation and perfusion distribution in intubated patients on VA-ECMO

SUMMARY:
There is limited data on the respiratory system mechanics and ideal mode of ventilation for patients on veno-arterial extra-corporeal membrane oxygenation (VA ECMO) post cardiac arrest. In this observational study, the investigators will review and/or obtain laboratory, hemodynamic, respiratory system mechanical, and clinical data from patients on VA ECMO. The specific aims of this study are as follows:

Aim 1: To characterize the lung ventilation strategy employed in patients on VA ECMO and its success.

Aim 2: To characterize respiratory system mechanics while on ECMO using esophageal manometry and Electrical Impedance Tomography (EIT).

Aim 3: To characterize right heart function and pulmonary vascular hemodynamics on the employed ventilation strategy.

The overarching hypothesis is that fine-tuned individualized ventilation might be superior to an algorithm that does not account for cardiac and pulmonary functions. Therefore, the aims of this study are to identify areas in which the ventilation strategy may theoretically be suboptimal, which will guide future interventional studies investigating alternatives methods of ventilation which may reduce time on the ventilator after cardiac arrest, time in the intensive care unit, and need for veno-venous ECMO.

ELIGIBILITY:
Inclusion Criteria:

* On VA ECMO after cardiac arrest
* Between 18 and 85 years of age
* Has an orogastric or nasogastric tube with esophageal balloon capabilities in place

Exclusion Criteria:

* Known pre-existing significant pulmonary pathology
* Pacemaker or implanted cardiac defibrillator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients without underlying pulmonary disease on VA ECMO post-cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-01-09 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Percent of total distribution of ventilation by region, on given ventilator settings | Within 24-48 hours of ECMO cannulation
  EIT will be used to determine the percent of total ventilation occurring in each of four lung quadrants on an axial plane: right upper, left upper, right lower, and left lower.

SECONDARY OUTCOMES:
Time on VA-ECMO | 14 days, 90 days
Need to transition to VV-ECMO | 14 days, 90 days
Time on mechanical ventilation | 14 days, 90 days
Time in ICU | 14 days, 90 days
90-day mortality | 90 days
Incidence of ventilator-associated pneumonia | 14 days, 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided